CLINICAL TRIAL: NCT04316676
Title: MyocardiAl CT Perfusion and Coronary Flow: a CompreHensive Cardiac CT Myocardial Perfusion Imaging (MPI)/Fractional Flow Reserve (FFR) and PET-CT MPI Evaluation (The MATCH Investigation)
Brief Title: The MATCH Investigation: CT Myocardial Perfusion and CT-FFR vs PET MPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Carlo N. De Cecco, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00114434
Record Dates: First submitted 2020-03-16; First posted 2020-03-20 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Atherosclerosis; Cardiovascular disease; Myocardial ischemia; Imaging; Nuclear medicine; Radiology
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Cardiovascular Diseases; Myocardial Ischemia | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Three imaging techniques: PET-MPI, CT-MPI, and CT-FFR (Other): Participants referred for a clinical PET-MPI will also have CT-MPI and CT-FFR imaging performed for analysis of myocardial perfusion.
  Interventions: Diagnostic Test: PET-MPI Protocol; Diagnostic Test: CT-MPI; Diagnostic Test: Coronary CT angiography (CCTA) for CT-FFR calculation; Drug: Regadenoson

INTERVENTIONS:
Diagnostic Test: PET-MPI Protocol — Patients with suspected CAD who are referred to a clinical PET-MPI will undergo the standard clinical protocol applied in the Emory Nuclear Medicine department.
Diagnostic Test: CT-MPI — For the CT-MPI, dynamic volume CT myocardial perfusion applying the "dynamic shuttle" mode will be used to rapidly cover the entire cardiac anatomy during infusion of a contrast medium bolus for monitoring bolus passage through the left ventricular myocardium. The "dynamic shuttle" mode consists of an image acquisition during rapid, yet smooth back-and-forth movement of the CT scanner table, so that contrast media bolus passage can be evaluated within the entire left ventricle in a time-resolved fashion. This scan acquisition will be performed during pharmacologically induced stress and during rest conditions. CT-MPI studies will be contrast medium enhanced by 50-70 ml of iodinated contrast agent, administered at a flow rate of 5 mL/s. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
Diagnostic Test: Coronary CT angiography (CCTA) for CT-FFR calculation — Coronary CT angiography (CCTA) will be performed for delineation of the coronary arteries, detection of potential coronary stenosis and FFR calculation. CCTA will be performed at rest following administration of intravenous contrast agent (50-70 mL of iodinated contrast material at a flow rate of 4-5 mL/s). A total radiation dose of approximately 8 millisievert (mSv) has expected to be administered with the stress/rest protocol to the patient. The total amount of contrast agent will not exceed 140 ml. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
Drug: Regadenoson — Pharmacological stress testing for the CT-MPI scan will be performed with a single injection of 0.4 mg of regadenoson (Lexiscan).
  Other Names: Lexiscan

SUMMARY:
The overall goal of this project is to compare the absolute quantification of myocardial perfusion done by using CT myocardial perfusion imaging (CT-MPI) and the coronary flow measured by using CT Fractional Flow Reserve analysis (CT-FFR) to the gold standard represented by PET myocardial perfusion imaging (PET-MPI).

DETAILED DESCRIPTION:
Participants will be patients who are scheduled to undergo PET Myocardial Perfusion Imaging, which is the traditional method for evaluating patients with suspected blockages or narrowing of the heart vessels (coronary artery disease) causing impaired blood to flow to the heart muscle (myocardium).

The purpose of the study is to determine and compare the newest heart imaging equipment which allows the non-invasive evaluation of coronary anatomy, coronary flow and myocardial perfusion in patients with suspected or proven coronary artery disease (CAD) with the actual gold-standard for quantitative myocardial perfusion assessment. In order to achieve this aim, the study team will compare heart scan results from a computed tomography (CT) Myocardial Perfusion Imaging (CT-MPI) scan and CT-Fractional Flow Reserve (FFR) with the actual standard clinical care represented by a PET Myocardial Perfusion Imaging (PET-MPI) study.

ELIGIBILITY:
Inclusion Criteria:

* Referred for a clinically indicated CT-MPI for CAD assessment
* Must provide written informed consent prior to any study-related procedures being performed
* Must be willing to comply with all clinical study procedures

Exclusion Criteria:

* Pregnant or nursing females. The possibility of pregnancy will be excluded by testing (serum or urine ßHCG) within 24 hours before study agent administration, or if the woman has previous surgical sterilization, or if the woman is post-menopausal, with minimum one (1) year history without menses.
* Currently taking or has taken within 48 hours the following excluded medications:

  * ActoPlus Met (Pioglitazone + metformin)
  * Avandamet (Rosiglitazone + metformin)
  * Fortamet (metformin)
  * Glucovance (Glyburide +metformin)
  * Glucophage (metformin)
  * Glucophage extended-release (XR) (metformin)
  * Glumetza (metformin)
  * Janumet (Sitagliptin + metformin)
  * Metformin
  * Metaglip (Glipizide + metformin)
  * Riomet (metformin)
* Acute psychiatric disorder
* Unwilling to comply with the requirements of the protocol
* Previously entered this study
* Known hypersensitivity to iodinated contrast material, beta-blockers, or pharmaceutical stressors used in this study
* Suffers from claustrophobia
* Impaired renal function (GFR < 45 ml/min)
* Acute hypotension (<100 mm Hg systolic)
* 2nd or 3rd degree atrioventricular (AV) block

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo De Cecco, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital in Atlanta, Georgia, USA. Participant enrollment began June 16, 2021 and all follow-up assessments were completed by September 24, 2024.
Groups:
- Three Imaging Techniques: PET-MPI, CT-MPI, and CCTA for CT-FFR Calculation: Participants referred for a clinical positron emission tomography myocardial perfusion imaging (PET-MPI), the gold standard for evaluating patients with suspected coronary blockages or coronary artery disease, also attend a study visit where they have computed tomography (CT) myocardial perfusion imaging (CT-MPI) and coronary CT angiography for calculation of CT fractional flow reserve (CT-FFR) imaging performed for analysis of myocardial perfusion. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
Period: Overall Study
Arm/Group | Three Imaging Techniques: PET-MPI, CT-MPI, and CCTA for CT-FFR Calculation
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Three Imaging Techniques: PET-MPI, CT-MPI, and CT-FFR: Participants referred for a clinical positron emission tomography myocardial perfusion imaging (PET-MPI), the gold standard for evaluating patients with suspected coronary blockages or coronary artery disease, also attend a study visit where they have computed tomography (CT) myocardial perfusion imaging (CT-MPI) and coronary CT angiography for calculation of CT fractional flow reserve (CT-FFR) imaging performed for analysis of myocardial perfusion. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
Arm/Group | Three Imaging Techniques: PET-MPI, CT-MPI, and CT-FFR
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated as weight in kilograms (kg) / height in meters (m)^2
  kg/m^2 | 34.9 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Blood Flow
Description: The absolute quantification of myocardial perfusion between CT-MPI and PET-MPI is compared. Myocardial perfusion is quantified using appropriate tracer kinetic models resulting myocardial blood flow mL/g/min.
Time Frame: Day of PET-MPI Scan, and Day of CT-MPI and CT-FFR Scans (up to 90 days)
Population: PET-MPI data were lost for two participants during an equipment move.
Measure: Mean (Standard Deviation); unit: mL/g/min
Groups:
- CT-MPI: Participants referred for a clinical positron emission tomography myocardial perfusion imaging (PET-MPI), the gold standard for evaluating patients with suspected coronary blockages or coronary artery disease, also attend a study visit where they have computed tomography (CT) myocardial perfusion imaging (CT-MPI) and coronary CT angiography for calculation of CT fractional flow reserve (CT-FFR) imaging performed for analysis of myocardial perfusion. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
  For the CT-MPI, dynamic volume CT myocardial perfusion applying the "dynamic shuttle" mode is used to rapidly cover the entire cardiac anatomy during infusion of a contrast medium bolus for monitoring bolus passage through the left ventricular myocardium. This scan acquisition is performed during pharmacologically induced stress and during rest conditions. CT-MPI studies are contrast medium enhanced by an iodinated contrast agent. Pharmacological stress testing for the CT-MPI scan is performed with a single injection of 0.4 mg of regadenoson.
- PET-MPI - Rest: Participants referred for a clinical positron emission tomography myocardial perfusion imaging (PET-MPI), the gold standard for evaluating patients with suspected coronary blockages or coronary artery disease (CAD), also attend a study visit where they have computed tomography (CT) myocardial perfusion imaging (CT-MPI) and coronary CT angiography for calculation of CT fractional flow reserve (CT-FFR) imaging performed for analysis of myocardial perfusion. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
  Patients with suspected CAD who are referred to a clinical PET-MPI undergo the standard clinical protocol applied in the Emory Nuclear Medicine department. PET-MPI is performed with stress and rest conditions.
- PET-MPI - Stress: Participants referred for a clinical positron emission tomography myocardial perfusion imaging (PET-MPI), the gold standard for evaluating patients with suspected coronary blockages or coronary artery disease, also attend a study visit where they have computed tomography (CT) myocardial perfusion imaging (CT-MPI) and coronary CT angiography for calculation of CT fractional flow reserve (CT-FFR) imaging performed for analysis of myocardial perfusion. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
  Patients with suspected CAD who are referred to a clinical PET-MPI undergo the standard clinical protocol applied in the Emory Nuclear Medicine department. PET-MPI is performed with stress and rest conditions.
Arm/Group | CT-MPI | PET-MPI - Rest | PET-MPI - Stress
Number analyzed (Participants) | 20 | 18 | 18
mL/g/min | 1.60 (0.43) | 0.96 (0.29) | 2.40 (1.09)

2. Primary Outcome: Coronary Flow Per CT-FFR
Description: Coronary flow is measured using the CT-FFR calculation with the CCTA scans. CT-FFR measures blood flow through coronary arteries and is used clinically to quantify the severity of CAD to determine further interventions. CT-FFR is the ratio between the blood flow (BF) in a diseased artery and a normal artery. Clinically, the CT-FFR calculation is only useful in patients with intermediate stenosis because stenosis below intermediate results in a value that is near zero and the calculation cannot be performed when stenosis is complete. The normal range for CT-FFR is greater than 0.80, values of 0.76 to 0.80 are borderline while values of 0.75 or less are associated with a high likelihood of reduced blood flow (ischemia).
Time Frame: Day of CT-MPI and CCTA scans
Population: Only one participant met clinical guidelines for the calculation of CT-FFR by having intermediate stenosis. One participant had stenosis too high to calculate CT-FFR while the remaining 18 participants had too little stenosis for an informative calculation.
Measure: Number; unit: ratio
Groups:
- Coronary CT Angiography (CCTA) for CT-FFR Calculation: Participants referred for a clinical positron emission tomography myocardial perfusion imaging (PET-MPI), the gold standard for evaluating patients with suspected coronary blockages or coronary artery disease, also attend a study visit where they have computed tomography (CT) myocardial perfusion imaging (CT-MPI) and coronary CT angiography for calculation of CT fractional flow reserve (CT-FFR) imaging performed for analysis of myocardial perfusion. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
  Coronary CT angiography (CCTA) is performed for delineation of the coronary arteries, detection of potential coronary stenosis and fractional flow reserve (FFR) calculation. CCTA is performed at rest following administration of intravenous contrast agent.
Arm/Group | Coronary CT Angiography (CCTA) for CT-FFR Calculation
Number analyzed (Participants) | 1
ratio | 1.29

3. Primary Outcome: Sensitivity of Myocardial Perfusion Abnormalities Diagnosis
Description: The accuracy of detection of myocardial perfusion abnormalities is compared between PET-MPI, CT-MPI, CCTA, and CT-FFR approach. Diagnostic accuracy using CT-MPI, CCTA and CT-FFR is calculated as sensitivity (true positives) with PET as the reference standard.
Time Frame: Day 1 (day of scans)
Population: This analysis includes participants with a PET-MPI result available. PET-MPI data were lost for two participants during an equipment move. Only one participant met clinical guidelines for the calculation of CT-FFR by having intermediate stenosis, however, the gold standard PET exam provided an incorrect diagnosis thus calculating sensitivity cannot correctly estimate the accuracy of CT-FFR.
Measure: Number; unit: percentage of true postive cases
Groups:
- CCTA with CT-FFR Calculation: Participants referred for a clinical positron emission tomography myocardial perfusion imaging (PET-MPI), the gold standard for evaluating patients with suspected coronary blockages or coronary artery disease, also attend a study visit where they have computed tomography (CT) myocardial perfusion imaging (CT-MPI) and coronary CT angiography for calculation of CT fractional flow reserve (CT-FFR) imaging performed for analysis of myocardial perfusion. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
  Coronary CT angiography (CCTA) is performed for delineation of the coronary arteries, detection of potential coronary stenosis and fractional flow reserve (FFR) calculation. CCTA is performed at rest following administration of intravenous contrast agent.
- CCTA: Participants referred for a clinical positron emission tomography myocardial perfusion imaging (PET-MPI), the gold standard for evaluating patients with suspected coronary blockages or coronary artery disease, also attend a study visit where they have computed tomography (CT) myocardial perfusion imaging (CT-MPI) and coronary CT angiography for calculation of CT fractional flow reserve (CT-FFR) imaging performed for analysis of myocardial perfusion. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
  Coronary CT angiography (CCTA) is performed for delineation of the coronary arteries and detection of potential coronary stenosis. CCTA is performed at rest following administration of intravenous contrast agent.
Arm/Group | CT-MPI | CCTA with CT-FFR Calculation | CCTA
Number analyzed (Participants) | 18 | 0 | 18
percentage of true postive cases | 100 |  | 100

4. Primary Outcome: Specificity of Myocardial Perfusion Abnormalities Diagnosis
Description: The accuracy of detection of myocardial perfusion abnormalities is compared between PET-MPI, CT-MPI, CCTA, and CT-FFR approach. Diagnostic accuracy using CT-MPI, CCTA and CT-FFR is calculated as specificity (true negatives) with PET as the reference standard.
Time Frame: Day 1 (day of scans)
Population: This analysis includes participants with a PET-MPI result available. PET-MPI data were lost for two participants during an equipment move. Only one participant met clinical guidelines for the calculation of CT-FFR by having intermediate stenosis, however, the gold standard PET exam provided an incorrect diagnosis thus calculating specificity cannot correctly estimate the accuracy of CT-FFR.
Measure: Number; unit: percentage of true negative cases
Arm/Group | CT-MPI | CCTA with CT-FFR Calculation | CCTA
Number analyzed (Participants) | 18 | 0 | 18
percentage of true negative cases | 100 |  | 94

5. Primary Outcome: Area Under the Curve (AUC) for Detection of Myocardial Perfusion Abnormalities
Description: The accuracy of detection of myocardial perfusion abnormalities is compared between PET-MPI, CT-MPI, CCTA, and CT-FFR approach. Diagnostic accuracy using CT-MPI, CCTA and CT-FFR is calculated as overall AUC with PET as the reference standard. The AUC examines the overall accuracy of a diagnostic test. Higher AUC indicates greater accuracy in detecting myocardial perfusion abnormalities with 1.0 being 100% accurate. An AUC value of 0.5 indicates that the test is as accurate as random chance.
Time Frame: Day 1 (day of scans)
Population: This analysis includes participants with a PET-MPI result available. PET-MPI data were lost for two participants during an equipment move.
Measure: Number; unit: probabliity of accurate detection
Arm/Group | CT-MPI | CCTA with CT-FFR Calculation | CCTA
Number analyzed (Participants) | 18 | 1 | 18
probabliity of accurate detection | 1.00 | 0 | 0.97

6. Primary Outcome: Sensitivity of Coronary Stenosis Diagnosis
Description: The accuracy of detection of coronary stenosis is compared between PET-MPI, CT-MPI, and CCTA with CT-FFR approach. Diagnostic accuracy is calculated as sensitivity (true positives) with CCTA as the reference standard.
Time Frame: Day 1 (day of scans)
Population: as for outcome 5
Measure: Number; unit: percentage of true postive cases
Groups:
- PET-MPI: Participants referred for a clinical positron emission tomography myocardial perfusion imaging (PET-MPI), the gold standard for evaluating patients with suspected coronary blockages or coronary artery disease, also attend a study visit where they have computed tomography (CT) myocardial perfusion imaging (CT-MPI) and coronary CT angiography for calculation of CT fractional flow reserve (CT-FFR) imaging performed for analysis of myocardial perfusion. The CT examinations are scheduled within 90 days of the standard clinical PET examination.
  Patients with suspected CAD who are referred to a clinical PET-MPI undergo the standard clinical protocol applied in the Emory Nuclear Medicine department. PET-MPI is performed at rest and with stress.
Arm/Group | CT-MPI | PET-MPI | CCTA with CT-FFR Calculation
Number analyzed (Participants) | 18 | 18 | 1
percentage of true postive cases | 67 | 67 | 100

7. Primary Outcome: Specificity of Coronary Stenosis Detection
Description: The accuracy of detection of coronary stenosis is compared between PET-MPI, CT-MPI, and CCTA with CT-FFR approach. Diagnostic accuracy is calculated as specificity (true negatives) with CCTA as the reference standard.
Time Frame: Day 1 (day of scans)
Population: This analysis includes participants with a PET-MPI result available. PET-MPI data were lost for two participants during an equipment move. Specificity could not be calculated in the CCTA with CT-FFR Calculation study arm as there was not a participant negative for coronary stenosis per the reference standard.
Measure: Number; unit: percentage of true negative cases
Arm/Group | CT-MPI | PET-MPI | CCTA with CT-FFR Calculation
Number analyzed (Participants) | 18 | 18 | 0
percentage of true negative cases | 100 | 100 |

8. Primary Outcome: Area Under the Curve for Detection of Coronary Stenosis
Description: The accuracy of detection of coronary stenosis is compared between PET-MPI, CT-MPI, and CCTA with CT-FFR approach. Diagnostic accuracy is calculated as overall AUC with CCTA as the reference standard. The AUC examines the overall accuracy of a diagnostic test. Higher AUC indicates greater accuracy in detecting coronary stenosis with 1.0 being 100% accurate. An AUC value of 0.5 indicates that the test is as accurate as random chance.
Time Frame: Day 1 (day of scans)
Population: as for outcome 5
Measure: Number; unit: probabliity of accurate detection
Arm/Group | CT-MPI | PET-MPI | CCTA with CT-FFR Calculation
Number analyzed (Participants) | 18 | 18 | 1
probabliity of accurate detection | 0.83 | 0.83 | 1

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected during the PET-MPI scan and during the CT-MPI and CCTA scans, for a total of two days spread over a period of up to 90 days.
Arm/Group | PET-MPI | CT-MPI | CCTA With CT-FFR Calculation
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT04316676/Prot_SAP_000.pdf